CLINICAL TRIAL: NCT04063553
Title: Impact of Volunteerism in the Acute Setting: Guiding Rehabilitative Exercises in Patients After Total Knee Replacement (TKR). A Pilot Study
Brief Title: Impact of Volunteerism in the Acute Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Eng Chan Neoh, Senior Physiotherapist, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018/00638
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled trial, eligible subjects will be randomised by research coordinator to either control or intervention group based on block randomisation with sealed envelop.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will be blinded from the group allocation. Research coordinator will be the the only person handling randomization, group allocation, arrange for volunteers to attend to the patient or not, and arrange for assessor to assess the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Other): Subjects in the intervention group will receive standard physiotherapy care and an additional volunteers session once a day for at least 3 times during their stay in the hospital. The volunteer will set up the TKR exercise video for the subjects, then supervise or guide the subjects with the exercises.
  Interventions: Other: Volunteers Service
- Control arm (Other): The control group subjects will receive only standard physiotherapy care and they will be instructed to perform 1 set of exercises daily following a brochure given
  Interventions: Other: Exercise brochure

INTERVENTIONS:
Other: Volunteers Service — Subjects in the intervention group will receive standard physiotherapy care and an additional volunteers session once a day for at least 3 times during their stay in the hospital. The volunteer will set up the TKR exercise video for the subjects, then supervise or guide the subjects with the exercises.
  All volunteers are recruited from TTSH volunteers pool managed by Center of Health Activation (CHA). TKR volunteers are trained by the study team, including a formal classroom session and a practical and role play session. After the training, volunteers need to pass 3 assessment by the physiotherapists in order to attend to patients independently by themselves. Volunteers who are bilingual will attend to the subject alone, or else those who can only converse in Chinese/ English will pair up with another volunteer who knows another language to make sure there is no communication barrier between volunteers and patients.
  Arms: Intervention arm
Other: Exercise brochure — . The control group subjects will receive only standard physiotherapy care and they will be instructed to perform 1 set of exercises daily following a brochure given. The exercises in the brochure and exercises taught by the volunteers are the same. The video and brochure are available in both English and Chinese version.
  Arms: Control arm

SUMMARY:
Rehabilitation, with a particular emphasis on physiotherapy and exercise, is widely promoted and strongly recommended after total knee replacement (TKR). The primary goals of rehabilitation are to improve knee range-of-motion, muscle strength, functional mobility and perceived quality of life. Exercises are usually prescribed and guided by a physiotherapist attending to the patient. The intensity of rehabilitation has an impact on clinical outcome. A study done by Lee et al in 2012 concluded that higher exercise dose translates to better function after TKR, especially in older population and for those with higher pain. Various literatures has also strongly recommended twice a day rehabilitation session for patients after TKR (Cook et al, 2008; Smith et al 2012).

DETAILED DESCRIPTION:
Rehabilitation, with a particular emphasis on physiotherapy and exercise, is widely promoted and strongly recommended after total knee replacement (TKR). The primary goals of rehabilitation are to improve knee range-of-motion, muscle strength, functional mobility and perceived quality of life. Exercises are usually prescribed and guided by a physiotherapist attending to the patient. The intensity of rehabilitation has an impact on clinical outcome. A study done by Lee et al in 2012 concluded that higher exercise dose translates to better function after TKR, especially in older population and for those with higher pain. Various literatures has also strongly recommended twice a day rehabilitation session for patients after TKR (Cook et al, 2008; Smith et al 2012). The standard practice in the in-patient setting is that physiotherapist will attend to the TKR patients once a day and remind patients to perform exercises by themselves, following the exercise booklet given, during their free time in the ward to maximise their recovery. However, due to post-operative fatugue, pain and fearful of movement, most of the patients are not compliant to the exercises given.

Volunteers have been present in health care settings for centuries. Several studies have shown that volunteers can be an essential part of the healthcare system. They are commonly involved in non-clinical tasks such as providing emotional support to patients and families (Burbeck et al., 2014), assisting with meals (Robinson et al., 2014) and facilitating recreational activities in patients with dementia (Hall et al., 2017).

However, no study has investigated the involvement of volunteers in actual clinical work. Our study aim to explore the feasibility of volunteers involvement in teaching and guiding exercises which conventionally done by physiotherapists, and to investigate the effectiveness of such volunteer service. There is no existing evidence on volunteers dealing with elderly patients in acute stage right after surgery as well, and this clinical research will be the first to explore that.

ELIGIBILITY:
Inclusion Criteria:

* Standard unilateral TKR without complications
* 55 years or older
* Pain less than or equal to 6/10 (i.e or between mild to moderate)
* Cognitively intact (able to follow at least 1-step instruction consistently)
* Vitals stable (Blood pressure, HR, oxygen saturation)
* Able to verbalise understanding and give informed consent
* Able to understand Mandarin or English

Exclusion Criteria:

* Unable to follow instructions consistently due to
* Cognitive impairment (Dementia, delirium)
* Behavioural issues (Confused, aggressive)
* Visually or hearing impaired
* Language illiteracy (listening)
* Medically unstable such as Hb drop (< 8) , acute desaturation
* Reduced exercises tolerance- Unable to tolerate a 20 minutes exercise session
* Post-operative complication such as delirium, DVT, cardiac issues.
* Excessive bleeding from the wound dressing

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Knee flexion and extension range of motion | through study completion, an average of 5 days
  knee range of motion will be measured using goniometer
Quadriceps strength | through study completion, an average of 5 days
  Quads strength will be assessed by using handheld dynamo-meter

SECONDARY OUTCOMES:
Pain intensity | through study completion, an average of 5 days
  pain intensity will be assessed by using VAS scale. VAS scale is a valid scale to assess pain intensity. It is a likert scale with 0-10 with 0 is no pain and 10 is maximum pain, Subject will be asked to give a number based on the pain level that they feel.
Timed up and Go test | through study completion, an average of 5 days
  Functional test to measure the duration needed to complete the task
Length of stay | through study completion, an average of 5 days
  Length of hospital stay to discharge home
survey | through study completion, an average of 5 days
  survey with likert scale 1-5 to investigate patient acceptance and satisfaction level towards volunteer service
quiz | through study completion, an average of 5 days
  quiz with Yes or No to test the knowledge of subjects about post TKR rehab

CONTACTS AND LOCATIONS:
Overall Officials: Eng Chuan Neoh, masters, Principal Investigator — Senior Physiotherapist
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No